CLINICAL TRIAL: NCT06539117
Title: Early Initiation of Oral Feeding Versus Traditional Feeding Post Caesarean Section: A Randomized Controlled Trial
Brief Title: Early Initiation of Oral Feeding Versus Traditional Feeding Post Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Darlington-Peter Chibuzor Ugoji (Other)
Responsible Party: Sponsor-Investigator, Darlington-Peter Chibuzor Ugoji, Principal Investigator, Alex Ekwueme Federal University Teaching Hospital
Organization: Alex Ekwueme Federal University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NHREC/16/05/22/185
Record Dates: First submitted 2024-04-14; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Complication; Postoperative
Keywords: Caesarean section; Post-operative feeding; Paralytic ileus
MeSH Terms: conditions — Intestinal Pseudo-Obstruction

STUDY DESIGN:
Intervention Model Description: Open labeled equivalence randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EARLY FEEDING GROUP (Experimental): In this group, participants were encouraged to commence oral sips of 150 millilitres of water from 6 hours post-caesarean delivery by the staff nurse. Thereafter, they were given semi-solid diet (250 milliliter of pap) from the 12th hour, and subsequently solid diet (a plate of well- cooked rice) by the trained nursing staff.
  Interventions: Other: Early feeding post caesarean section
- TRADITIONAL FEEDING GROUP (Active Comparator): Participants in this group were managed traditionally by restricting commencement of oral fluid intake until after 24 hours. They were allowed intake of oral sips of 150 millilitres of water after 24 hours post-caesarean section, thereafter, 250 millilitres of pap and subsequently solid diet (a plate of well-cooked rice)
  Interventions: Other: Early feeding post caesarean section

INTERVENTIONS:
Other: Early feeding post caesarean section — In this group, participants were encouraged to commence oral sips of 150 millilitres of water from 6 hours post-caesarean delivery by the staff nurse. Thereafter, they were given semi-solid diet (250 milliliter of pap) from the 12th hour, and subsequently solid diet (a plate of well- cooked rice) by the trained nursing staff.

SUMMARY:
Early initiation of oral feeding, within 6-12 hours post-caesarean section, has been noticed to be well tolerated by patients and helps them recover fast. Our study aimed to evaluate the tolerability, safety and benefits of early oral feeding post-caesarean section.

DETAILED DESCRIPTION:
BACKGROUND: Early initiation of oral feeding, within 6-12 hours post-caesarean section, has been noticed to be well tolerated by patients and helps them recover fast. However, the traditional method of waiting for 24 hours to commence oral feeding post-caesarean section is still being widely practiced due to the fear of post-operative ileus. Though some studies have shown this fear to be unfounded, early initiation of oral feeding is not yet universally accepted.

OBJECTIVES: To evaluate the tolerability, safety and benefits of early oral feeding post-caesarean section.

STUDY DESIGN AND SETTING: This was a randomized control trial (equivalence) carried out at Alex Ekwueme Federal University Teaching Hospital Abakaliki, Nigeria.

METHODS: Three hundred and six eligible women, randomized into groups (A=early and B=traditional feeding group) were admitted into the post natal ward after elective or emergency caesarean section. Women in group A were commenced on graded oral sips 6 hours post- caesarean section and subsequently soft diets from the 12th hour, after oral sips were well tolerated, while those in group B were commenced on the same regimen as in group A 24 hours post-caesarean section.

MAIN OUTCOME MEASURE: Time of return of bowel sound, time of resuming normal diets, duration of hospital stay, and post-operative complications ANALYSIS: Data obtained were analyzed using the computer software, IBM SPSS version 26. Frequency tables were made and results tested for significance using the t-test for continuous variables and Chi-square test for categorical variables. Relative risk (RR) was also determined, with confidence interval set at 95% and the level of significance determined by p-value < 0.05

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women included in this study were those booked for elective or emergency caesarean section under spinal anaesthesia, for various indications from antenatal clinic, antenatal ward, labour ward and obstetric emergency unit who met inclusion criteria and consented to the study.

Exclusion Criteria:

* Women with prolonged obstructed labour.
* Women with immunosuppression or HIV/AIDS
* Women with eclampsia.
* Women with medical complications of pregnancy such as:
* Sickle cell anaemia, uncontrolled diabetes, uncontrolled hypertension.
* Women who received general anaesthesia
* Women with previous history of bowel surgery
* Women on drugs that can cause constipation
* Women with previous history of chronic constipation

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Post Caesarean section
Enrollment: 153 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Rate of tolerability of oral sips | 48hours
  This was the rate of tolerability of oral sips especially in the first 48 hours post surgery as shown by absence of complications such as nausea, vomiting, abdominal distention and paralytic ileus.

CONTACTS AND LOCATIONS:
Overall Officials: DARLINTON-PETER CHIBUZOR C UGOJI, MBBS, Principal Investigator — Alex Ekwueme Federal University Teaching Hospital
Locations (1):
- AEFUTHA, Abakaliki, Ebonyi State, Nigeria

IPD SHARING:
Plan to Share IPD: No
This will be following publication

REFERENCES:
- [Result] Mamah J.E, Asiegbu O, Asiegbu U, Nnadozie U, Okafor L. A six-year review of caesarean section at the Federal Teaching Hospital Abakaliki, Ebonyi State, South East Nigeria. Open Journal of Obstetrics and Gynaecology, 2020 Dec,11; (10) 1669-1676.